CLINICAL TRIAL: NCT02997306
Title: COEBICS: Comparison of Erythema Between Interrupted and Continuous Sutures
Acronym: COEBICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, David Zloty, Clinical Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H16-01802
Record Dates: First submitted 2016-12-07; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Surgical Scar Erythema
Keywords: Moh's Surgery; Erythema; Face; Simple Interrupted Sutures; Running Sutures; Image Processing
MeSH Terms: conditions — Erythema; Facies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Superior/Medial Running Sutures (Experimental): In this cohort, the running sutures will be randomized to be oriented on Superior/Medial half of the scar, and the remaining half of the scar will be closed with simple interrupted sutures.
  Interventions: Procedure: Superior/Medial Running Sutures
- Inferior/Lateral Running Sutures (Experimental): In this cohort, the running sutures will be randomized to be oriented on Inferior/Lateral half of the scar, and the remaining half of the scar will be closed with simple interrupted sutures.
  Interventions: Procedure: Inferior/Lateral Running Sutures

INTERVENTIONS:
Procedure: Superior/Medial Running Sutures — Simple interrupted stitches and running (continuous) stitches are the two most frequently used suturing techniques. The erythema secondary to these suturing techniques will be compared by utilizing them side-by-side for closure of post-Moh's surgical defect repair in each patient. This intervention consists of running sutures being used for closure of the Superior/Medial half of the incision, and interrupted sutures being used on the Inferior/Lateral half of the incision.
  Arms: Superior/Medial Running Sutures
Procedure: Inferior/Lateral Running Sutures — Simple interrupted stitches and running (continuous) stitches are the two most frequently used suturing techniques. The erythema secondary to these suturing techniques will be compared by utilizing them side-by-side for closure of post-Moh's surgical defect repair in each patient. This intervention consists of running sutures being used for closure of the Inferior/Lateral half of the incision, and interrupted sutures being used on the Superior/Medial half of the incision.
  Arms: Inferior/Lateral Running Sutures

SUMMARY:
This is a randomized, controlled, prospective study which relies on computer-assisted skin image processing of scar photographs, to establish whether simple interrupted or running sutures are associated with the greatest degree of erythema when used to repair surgical defects arising from Moh's micrographic surgery (MMS) of facial skin cancers. Furthermore, through the use of the customized software that the investigators have developed for this purpose, an effort will be made to better understand the evolution (including progression and subsequent regression) of erythema over time in these scars.

DETAILED DESCRIPTION:
Purpose: This is a randomized, controlled, prospective split-scar study which employs computer-assisted image processing to establish whether simple interrupted or running sutures cause the greatest degree of erythema in the surgical scars resulting from Moh's micrographic surgery (MMS), and to better understand the evolution (including progression and subsequent regression) of erythema over time in these scars.

Hypothesis: Based on the literature review and the clinical experience of the investigators, it is hypothesized that the quantified difference in persisting erythema that is caused by each suturing technique will be minimal and not statistically significant.

Justification: The cosmetic appearance of scars is an important concern for patients undergoing Moh's micrographic surgery (MMS), a specialized therapeutic procedure that is used for high risk skin cancers on the face. Many factors influence the aesthetics of a surgical scar; suturing technique is among the most significant. Simple interrupted stitches and running (continuous) stitches are the two most frequently used suturing techniques. Anecdotal opinions favor one technique over the other. Some authors consider simple interrupted stitches to be more time consuming but allows more precise wound approximation. Other surgeons feel running stitches decrease suture marks. A recent literature search looking at the influence of suturing technique on the cosmetic outcome of scars could not draw any conclusion as to which stitching method should be recommended for facial repair because of the lack of comparative studies. The need for prospective randomized trials in this field is required. Multiple scales have been reported in the literature which can be utilized for cosmetic assessment of healing surgical scars. Persistent scar erythema/dilated peri-scar telangiectasias are a relatively common finding associated with facial surgery and are included as a component in only one of the aforementioned scar evaluation scales. Furthermore, it is only the presence of erythema that is gauged by the scale, and not its intensity or area as these parameters would be challenging to objectively assess. To address this issue, the investigators have developed a software that is capable of quantifying the intensity and area involving erythema in scars. As such, this study has been designed to determine whether simple interrupted or running sutures would cause the greatest degree of erythema and to what extent (both in terms of intensity and area) in the resulting facial MMS scars.

Objectives:

1. To determine whether simple interrupted or running sutures cause the greatest degree of persistent erythema in the scars resulting from MMS facial defect repair.
2. To determine the percentage difference in the degree of persisting erythema (including intensity and area) caused by each suturing technique.
3. To quantitatively assess the evolution of erythema over time in simple interrupted and running sutures to better characterize its patterns of progression and subsequent regression.

Research Design: Prospective randomized controlled split-scar study.

Research Methods: Subjects will be recruited at the Dermatologic Surgery Centre at the VGH Skin Care Centre. They will be offered the option to participate in this study prior to beginning their MMS procedure. All patients/accompanying family members will have adequate time to read the protocol and consent document prior to entering the surgical area. All surgeries will be performed by an experienced dermatologic surgeon and/or an MMS Fellow. The same procedure will be followed for each patient. After ensuring that the length of the scar will be >4cm, patients will be randomized (using computer generated sealed envelope method) to epidermal suturing technique. Depending on randomization, either the superior/medial or inferior/lateral half of the scar will be sutured with running stitches, whereas the other half will be closed with interrupted stitches. All other aspects of the procedures, including post-operative wound care and follow-up, will be similar as those for patients who are not in the study. The subjects will be seen again for follow up at 1 week, 8 weeks, and 6 months following their procedure, which are regularly scheduled for all patients who undergo MMS as part of their ongoing oncologic evaluation and wound care. No additional follow up appointments will be scheduled specifically for the purpose of this study. During each follow up appointment, close-up photographs of the scars will be taken using preset aperture (14), shutter speed (1/60 seconds), and flash settings (+1/3 exposure compensation) on a Canon EOS Digital Rebel XT, CanonMR-14EX ring flash, and Canon EFS 60mmf/2.8 macro lens. All photographs will be taken in the same follow-up room under closely matched lighting parameters and camera angles. Following their final reassessment at 6 months, all interval photos will be processed using the customized software to quantify intensity and area of erythema for each visit.

Statistical analysis: Power calculations have been performed. To detect a difference of 10% in the degree of erythema between the two study arms, with a power of 80%, 100 patients will be recruited. The two study arms are paired since each patient's scar is split into two parts. Subsequently, comparative paired t-tests will be performed on the software-generated values of erythema intensity and area for simple interrupted and running sutures from each interval MMS scar photograph.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included only if the following conditions are all met:

1. The subject is 18 years of age or older.
2. The subject is presenting with a facial surgical defect after MMS that requires a repair resulting in a scar of more than 4 cm in length.
3. The subject is willing and capable of cooperating to the extent and degree required by the protocol.

Exclusion Criteria:

Subjects will be excluded if any of the following conditions are met:

1. The subject has a history of keloidal scarring.
2. The subject will require radiation therapy after surgery.
3. The subject is participating in another investigational drug or device study within 30 days of proposed study enrolment.
4. The subject is not able to fully understand the protocol and consent documents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Intensity of Scar Erythema | 1 week, 8 weeks, and 6 months post-operatively
  The degree of scar erythema post-operatively will be assessed in each half of each patient's scar by quantifying both the intensity and the surface area of erythema. This will be achieved digitally by employing the customized software developed by the investigators for this purpose.

CONTACTS AND LOCATIONS:
Overall Officials: David Zloty, MD, FRCPC, Principal Investigator — Department of Dermatology and Skin Science, University of British Columbia
Locations (1):
- Dermatologic Surgery Centre at the Vancouver General Hospital Skin Care Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chuang GS, Leach BC, Wheless L, Lang PG, Cook J. Preoperative expectations and values of patients undergoing Mohs micrographic surgery. Dermatol Surg. 2011 Mar;37(3):311-9. doi: 10.1111/j.1524-4725.2011.01878.x. Epub 2011 Feb 22. PMID 21342309
- [Background] McLean NR, Fyfe AH, Flint EF, Irvine BH, Calvert MH. Comparison of skin closure using continuous and interrupted nylon sutures. Br J Surg. 1980 Sep;67(9):633-5. doi: 10.1002/bjs.1800670908. PMID 7000234
- [Background] Moy LS. Management of acute wounds. Dermatol Clin. 1993 Oct;11(4):759-66. PMID 8222359
- [Background] Moy RL, Waldman B, Hein DW. A review of sutures and suturing techniques. J Dermatol Surg Oncol. 1992 Sep;18(9):785-95. doi: 10.1111/j.1524-4725.1992.tb03036.x. PMID 1512311
- [Background] Quinn JV, Drzewiecki AE, Stiell IG, Elmslie TJ. Appearance scales to measure cosmetic outcomes of healed lacerations. Am J Emerg Med. 1995 Mar;13(2):229-31. doi: 10.1016/0735-6757(95)90100-0. PMID 7893315
- [Background] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752
- [Background] Sclafani AP, Sclafani JA, Sclafani AM. Successes, revisions, and postoperative complications in 446 Mohs defect repairs. Facial Plast Surg. 2012 Jun;28(3):358-66. doi: 10.1055/s-0032-1312691. Epub 2012 Jun 21. PMID 22723239